CLINICAL TRIAL: NCT01139827
Title: Association Between Framingham Risk Score, hsCRP and Vascular Inflammation: Analysis With 18F-Fluorodeoxyglucose Positron Emission Tomography
Status: Completed | Type: Observational
Sponsor: Korea University Guro Hospital (Other)
Other Study IDs: PET(FRS-CRP)
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-02

CONDITIONS: Cardiovascular Risk
Keywords: atherosclerosis; inflammation; hsCRP; Framingham risk score; positron emission tomography; inflammation in FDG-PET
MeSH Terms: conditions — Atherosclerosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal: normal group has no diabetes.
- IGT: IGT group has impaired fasting glucose or impaired glucose tolerance.

SUMMARY:
Framingham risk score is well known screening tool that detect cardiovascular (CV) risk. But it is not suitable for CV risk in mild risk group. So 18F-fluorodeoxyglucose positron emission tomography (FDG-PET) is a new imaging technique for detecting vascular inflammation within atherosclerotic plaques and hsCRP is also arising detection tool of CV risk.

The investigators are examining this association in normal and impaired glucose tolerance patients groups.

DETAILED DESCRIPTION:
We examined vascular inflammation using FDG-PET scan in 178 subjects (Normal and impaired glucose tolerance groups). Vascular 18F-FDG uptake was measured as both the mean and maximum blood-normalized standardized uptake value (SUV), known as the target-to-background ratio (TBR). And We analyzed that the association with Framingham risk score, hs CRP and vascular inflammation by FDG-PET scan.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* a history of cardiovascular disease (myocardial infarction, unstable angina, stroke or cardiovascular revascularization)
* active inflammatory disease, recent active infection
* stage 2 hypertension (resting blood pressure, ≥ 160/100 mmHg)
* diabetes mellitus
* systemic disorders such as severe hepatic, renal, and hematologic diseases
* taking drugs known to interfere with vascular inflammation measured by FDG-PET.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The subjects underwent routine health checkups at Korea University Guro Hospital. Patients with DM or gestational diabetes were not included.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea university guro hospital, Seoul, South Korea